CLINICAL TRIAL: NCT01236573
Title: Phase I/II Study of Metastatic Melanoma Using Lymphodepleting Conditioning Followed by Infusion of Tumor Infiltrating Lymphocytes Genetically Engineered to Express IL-12
Brief Title: Cell Therapy for Metastatic Melanoma Using CD8 Enriched Tumor Infiltrating Lymphocytes
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Unexpected toxicities, likely due to TIL/IL-12 & low % of durable responses.
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Steven Rosenberg, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 110011; 11-C-0011
Record Dates: First submitted 2010-11-05; First posted 2010-11-08 (Estimated); Results first posted 2015-10-26 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-10

CONDITIONS: Skin Cancer; Metastatic Melanoma
Keywords: Gene Therapy; Immunotherapy; Adoptive Cell Therapy; Metastatic Melanoma
MeSH Terms: conditions — Skin Neoplasms; Melanoma | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (11):
- Group 1 - CD8 + TIL expressing IL-12 1x10^6 (Experimental): Phase 1. Patients will receive a nonmyeloablative but lymphocyte depleting preparative regimen consisting of cyclophosphamide and fludarabine followed by intravenous infusion of interleukin-12 (IL-12) gene-transduced tumor infiltrating lymphocytes (TIL).
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: IL-12 transduced TIL
- Group 2 - CD8 + TIL expressing IL-12 3x10^6 (Experimental): Phase 1. Patients will receive a nonmyeloablative but lymphocyte depleting preparative regimen consisting of cyclophosphamide and fludarabine followed by intravenous infusion of IL-12 gene-transduced TIL.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: IL-12 transduced TIL
- Group 3 - CD8 + TIL expressing IL-12 1x10^7 (Experimental): Phase 1. Patients will receive a nonmyeloablative but lymphocyte depleting preparative regimen consisting of cyclophosphamide and fludarabine followed by intravenous infusion of IL-12 gene-transduced TIL.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: IL-12 transduced TIL
- Group 4- CD8+TIL expressing IL-12 3x10^7 (Experimental): Phase 1. Patients will receive a nonmyeloablative but lymphocyte depleting preparative regimen consisting of cyclophosphamide and fludarabine followed by intravenous infusion of IL-12 gene-transduced TIL.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: IL-12 transduced TIL
- Group 5 - Bulk TIL expressing IL-12 1x10^7 (Experimental): Phase 1. Patients will receive a nonmyeloablative but lymphocyte depleting preparative regimen consisting of cyclophosphamide and fludarabine followed by intravenous infusion of IL-12 gene-transduced TIL.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: IL-12 transduced TIL
- Group 6 - Bulk TIL expressing IL-12 3x10^7 (Experimental): Phase 1. Patients will receive a nonmyeloablative but lymphocyte depleting preparative regimen consisting of cyclophosphamide and fludarabine followed by intravenous infusion of IL-12 gene-transduced TIL.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: IL-12 transduced TIL
- Group 7- Bulk TIL expressing IL-12 1x10^8 (Experimental): Phase 1. Patients will receive a nonmyeloablative but lymphocyte depleting preparative regimen consisting of cyclophosphamide and fludarabine followed by intravenous infusion of IL-12 gene-transduced TIL.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: IL-12 transduced TIL
- Group 8 - Bulk TIL expressing IL-12 3x10^8 (Experimental): Phase 1. Patients will receive a nonmyeloablative but lymphocyte depleting preparative regimen consisting of cyclophosphamide and fludarabine followed by intravenous infusion of IL-12 gene-transduced TIL.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: IL-12 transduced TIL
- Group 9 - Bulk TIL expressing IL-12 1x10^9 (Experimental): Phase 1. Patients will receive a nonmyeloablative but lymphocyte depleting preparative regimen consisting of cyclophosphamide and fludarabine followed by intravenous infusion of IL-12 gene-transduced TIL.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: IL-12 transduced TIL
- Group 10- Bulk TIL expressing IL12 3x10^9 (Experimental): Phase 1. Patients will receive a nonmyeloablative but lymphocyte depleting preparative regimen consisting of cyclophosphamide and fludarabine followed by intravenous infusion of IL-12 gene-transduced TIL.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: IL-12 transduced TIL
- Group 11 - Bulk TIL expressing MTD 1x10^9 (Phase 2) (Experimental): Maximum tolerated dose (MTD). Patients will receive a nonmyeloablative but lymphocyte depleting preparative regimen consisting of cyclophosphamide and fludarabine followed by intravenous infusion of IL-12 gene-transduced TIL.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: IL-12 transduced TIL

INTERVENTIONS:
Drug: Fludarabine — Fludarabine 25 mg/m^2/day intravenous piggyback (IVPB) daily over 30 minutes for 5 days.
Drug: Cyclophosphamide — Cyclophosphamide 60 mg/kg/day X 2 days intravenous (IV) in 250 ml dextrose 5% in water (D5W) over 1 hr.
Biological: IL-12 transduced TIL — On day 0 (one to four days after the last dose of fludarabine), cells will be infused intravenously (i.v.) on the Patient Care Unit over 20 to 30 minutes.

SUMMARY:
Background:

- One experimental treatment for certain types of cancer is cell therapy, which involves collecting lymphocytes (white blood cells) from a tumor, growing them in the laboratory in large numbers, and then modifying the cells with a gene (interleukin-12 (IL-12)) that stimulates the immune system to attack and destroy the cancer cells. Because this treatment is experimental, researchers are interested in determining the side effects and overall effectiveness of cell therapy using white blood cells modified with IL-12 as a treatment for aggressive cancer.

Objectives:

- To determine the safety and effectiveness of cell therapy using IL-12 modified tumor white blood cells to treat metastatic melanoma.

Eligibility:

- Individuals greater than or equal to 18 years of age and less than or equal to age 66 who have been diagnosed with metastatic melanoma.

Design:

* Participants will be screened with a medical history, physical examination, blood and urine tests, and imaging studies.
* Cells for treatment will be collected during tumor biopsy or surgery.
* Prior to the start of cell therapy, participants will have imaging procedures, heart and lung function tests, and blood and urine tests, as well as leukapheresis to collect additional white blood cells.
* For 5 days before the cell infusion, participants will be admitted for inpatient chemotherapy with cyclophosphamide and fludarabine to suppress the immune system in preparation for the cell therapy.
* Participants will receive the modified white blood cells as an infusion 1 to 4 days after the last dose of chemotherapy. The day after the infusion, participants will receive filgrastim to stimulate blood cell growth.
* Participants will remain as inpatients for at least 5 to 10 days to recover from the treatment, and will be followed regularly after the treatment to study side effects and general effectiveness.
* Participants who initially respond to treatment but have a relapse may have one additional treatment using the same procedure.

DETAILED DESCRIPTION:
Background:

* Interleukin-12 (IL-12) is an important immunostimulatory cytokine. We have constructed a retroviral vector that contains an inducible single chain IL-12 driven by an nuclear factor of activated T-cells (NFAT) responsive promoter which can be used to mediate transfer of this gene into anti-tumor lymphocytes. This construct enables the secretion of IL-12 following stimulation of the T cell receptor.
* Transduction of the IL-12 gene into mouse anti-tumor lymphocytes results in a profound increase in the ability of these lymphocytes to mediate tumor regression following administration to tumor bearing mice. These cells have a profound advantage in inducing anti-tumor responses because very few cells are needed and there is no requirement for the concomitant administration of interleukin-2 (IL-2) as is the case for conventional cell transfer immunotherapies.
* Based on these murine studies we have now constructed a similar retrovirus that contains an inducible human single chain IL-12 driven by an NFAT responsive promoter. This retrovirus can be used to transduce tumor infiltrating lymphocytes (TIL) suitable for the therapy of patients with metastatic melanoma.

Objectives:

Primary objectives:

* To evaluate the safety of the administration of IL-12 engineered TIL in patients receiving a non-myeloablative conditioning regimen.
* Determine if the administration of IL-12 engineered TIL to patients following a non-myeloablative but lymphoid depleting preparative regimen will result in clinical tumor regression in patients with metastatic cancer.

Secondary objective:

-Determine the in vivo survival of IL-12 gene-engineered cells.

Eligibility:

Patients who are 18 years of age or older must have:

* metastatic melanoma;
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1;

Design:

* TIL will be resected from metastatic deposits and grown in IL-2 using standard techniques.
* Prior to approval of amendment A, after about 2 weeks TIL will undergo cluster of differentiation 8 (CD8) enrichment on a Miltenyi column and then undergo a rapid expansion by exposure to Muromoanb-CD3) OKT-3 an IL-2 in the presence irradiated feeder cells. Four to five days later, transduction is initiated by addition of retroviral vector supernatant containing the IL-12 gene.

With approval of amendment A, TIL will not undergo CD8 enrichment. Starting with cohort 5, after initial growth, TIL undergo a rapid expansion by exposure to OKT-3 and IL-2 in the presence irradiated feeder cells. Four to five days later, transduction is initiated by addition of retroviral vector supernatant containing the IL-12 gene.

* Patients will receive a nonmyeloablative but lymphocyte depleting preparative regimen consisting of cyclophosphamide and fludarabine followed by intravenous infusion of IL-12 gene-transduced TIL. Cohorts of 3 patients each will receive increasing cell doses.
* Patients will undergo complete evaluation of tumor with physical examination, computed tomography (CT) of the chest, abdomen and pelvis and clinical laboratory evaluation four to six weeks after treatment. If the patient has stable disease (SD) or tumor shrinkage, repeat complete evaluations will be performed every 1-3 months. After the first year, patients continuing to respond will continue to be followed with this evaluation every 3-4 months until off study criteria are met.
* The study will be conducted using a Phase I/II optimal design. The protocol will proceed in a phase 1 dose escalation design.
* Prior to approval of amendment A, the protocol enrolled 1 patient in each of the first 3 dose cohorts. Cohort 4 proceeded in a phase 1 dose escalation design, with of n=3. Should a single patient experience a dose limiting toxicity due to the cell transfer at a particular dose level, additional patients would be treated at that dose to confirm that no greater than 1/6 patients have a dose-limiting toxicity (DLT) prior to proceeding to the next higher level. If a level with 2 or more DLTs in 3-6 patients has been identified, three additional patients will be accrued at the next- lowest dose, for a total of 6, in order to further characterize the safety of the maximum tolerated dose.
* With approval of amendment A, no additional patients will be enrolled in cohort 4, and the protocol will enroll 1 patient in cohort 5 with a dose of 1 X 10^7 bulk young TIL cells. Cohorts 6-12 will proceeded in a phase 1 dose escalation design, with an n=3. Should a single patient experience a dose limiting toxicity due to the cell transfer at a particular dose level, additional patients would be treated at that dose to confirm that no greater than 1/6 patients have a DLT prior to proceeding to the next higher level. If a level with 2 or more DLTs in 3-6 patients has been identified, three additional patients will be accrued at the next-lowest dose, for a total of 6, in order to further characterize the safety of the maximum tolerated dose prior to starting the pahse II portion. If a dose limiting toxicity occurs in the cohort 4, that cohort will be expanded to 6 patients. If 2 DLTs are encountered in this cohort, the study will be terminated.
* Once the maximum tolerated dose (MTD) has been determined, the study then would proceed to the phase II portion using a phase II optimal design where initially 21 evaluable patients will be enrolled. If 0 or 1 of the 21 patients experiences a clinical response, then no further patients will be enrolled but if 2 or more of the first 21 evaluable patients enrolled have a clinical response, then accrual will continue until a total of 41 evaluable patients have been enrolled.
* The objective will be to determine if the combination of lymphocyte depleting chemotherapy, and IL-12 gene engineered lymphocytes is associated with a clinical response rate that can rule out 5% (p0=0.05) in favor of a modest 20% partial response (PR) + complete response (CR) rate (p1=0.20).

ELIGIBILITY:
* INCLUSION CRITERIA:
* Metastatic melanoma with evaluable disease.
* Greater than or equal to 18 years of age and less than or equal to age 66.
* Willing to sign a durable power of attorney
* Able to understand and sign the Informed Consent Document
* Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0 or 1
* Life expectancy of greater than three months
* Patients of both genders must be willing to practice birth control from the time of enrollment on this study and for up to four months after the cells are no longer detected in the blood.
* Serology:

  * Seronegative for human immunodeficiency virus (HIV) antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune-competence and thus be less responsive to the experimental treatment and more susceptible to its toxicities.)
  * Seronegative for hepatitis B antigen, and seronegative for hepatitis C antibody. If hepatitis C antibody test is positive, then patient must be tested for the presence of antigen by reverse transcription polymerase chain reaction (RT-PCR) and be hepatitis C virus ribonucleic acid (HCV RNA) negative.
  * Women of child-bearing potential must have a negative pregnancy test because of the potentially dangerous effects of the preparative chemotherapy on the fetus.
* Hematology:

  * Absolute neutrophil count greater than 1000/mm^3 without the support of filgrastim.
  * White blood cell (WBC) (> 3000/mm^3).
  * Platelet count greater than 100,000/mm^3.
  * Hemoglobin greater than 8.0 g/dl.
* Chemistry:

  * Serum alanine transaminase (ALT)/aspartate transaminase (AST) less or equal to 2.5 times the upper limit of normal.
  * Serum creatinine less than or equal to 1.6 mg/dl.
  * Total bilirubin less than or equal to 1.5 mg/dl, except in patients with Gilberts Syndrome who must have a total bilirubin less than 3.0 mg/dl.
* More than four weeks must have elapsed since any prior systemic therapy at the time the patient receives the preparative regimen, and patients toxicities must have recovered to a grade 1 or less (except for toxicities such as alopecia or vitiligo).

EXCLUSION CRITERIA:

* Previous treatment with interleukin-12 (IL-12).
* Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant.
* Active systemic infections, coagulation disorders or other major medical illnesses of the cardiovascular, respiratory or immune system, myocardial infarction, cardiac arrhythmias, obstructive or restrictive pulmonary disease.
* Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
* Concurrent opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities).
* Concurrent systemic steroid therapy.
* History of severe immediate hypersensitivity reaction to any of the agents used in this study.
* In patients > 60 years old and/or history of coronary revasularization or ischemic symptoms, documented left ventricular ejection fraction (LVEF) of less than or equal to 45%.

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Rosenberg, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Jemal A, Siegel R, Ward E, Murray T, Xu J, Thun MJ. Cancer statistics, 2007. CA Cancer J Clin. 2007 Jan-Feb;57(1):43-66. doi: 10.3322/canjclin.57.1.43. PMID 17237035
- [Background] Atkins MB, Lotze MT, Dutcher JP, Fisher RI, Weiss G, Margolin K, Abrams J, Sznol M, Parkinson D, Hawkins M, Paradise C, Kunkel L, Rosenberg SA. High-dose recombinant interleukin 2 therapy for patients with metastatic melanoma: analysis of 270 patients treated between 1985 and 1993. J Clin Oncol. 1999 Jul;17(7):2105-16. doi: 10.1200/JCO.1999.17.7.2105. PMID 10561265
- [Background] Gogas HJ, Kirkwood JM, Sondak VK. Chemotherapy for metastatic melanoma: time for a change? Cancer. 2007 Feb 1;109(3):455-64. doi: 10.1002/cncr.22427. PMID 17200963
- [Result] Zhang L, Morgan RA, Beane JD, Zheng Z, Dudley ME, Kassim SH, Nahvi AV, Ngo LT, Sherry RM, Phan GQ, Hughes MS, Kammula US, Feldman SA, Toomey MA, Kerkar SP, Restifo NP, Yang JC, Rosenberg SA. Tumor-infiltrating lymphocytes genetically engineered with an inducible gene encoding interleukin-12 for the immunotherapy of metastatic melanoma. Clin Cancer Res. 2015 May 15;21(10):2278-88. doi: 10.1158/1078-0432.CCR-14-2085. Epub 2015 Feb 18. PMID 25695689
- [Derived] Kerkar SP, Goldszmid RS, Muranski P, Chinnasamy D, Yu Z, Reger RN, Leonardi AJ, Morgan RA, Wang E, Marincola FM, Trinchieri G, Rosenberg SA, Restifo NP. IL-12 triggers a programmatic change in dysfunctional myeloid-derived cells within mouse tumors. J Clin Invest. 2011 Dec;121(12):4746-57. doi: 10.1172/JCI58814. Epub 2011 Nov 7. PMID 22056381

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1 - CD8 + TIL Expressing IL-12 1x10^6 (Phase 1); Group 2 - CD8 + TIL Expressing IL-12 3x10^6 (Phase 1); Group 3 - CD8 + TIL Expressing IL-12 1x10^7 (Phase 1); Group 4 - CD8 + TIL Expressing IL-12 3x10^7 (Phase 1); Group 5 - Bulk TIL Expressing IL-12 1x10^7 (Phase 1); Group 6 - Bulk TIL Expressing IL-12 3x10^7 (Phase 1); Group 7- Bulk TIL Expressing IL-12 1x10^8 (Phase 1); Group 8 - Bulk TIL Expressing IL-12 3x10^8 (Phase 1); Group 9 - Bulk TIL Expressing IL-12 1x10^9 (Phase 1); Group 10 - Bulk TIL Expressing IL12 3x10^9 (Phase 1); Group 11 - Bulk TIL Expressing MTD 1x10^9 (Phase 2): Patients will receive a nonmyeloablative but lymphocyte depleting preparative regimen consisting of cyclophosphamide and fludarabine followed by intravenous infusion of IL-12 gene-transduced TIL.
  Fludarabine: Fludarabine 25 mg/m2/day IVPB daily over 30 minutes for 5 days.
  Cyclophosphamide: Cyclophosphamide 60 mg/kg/day X 2 days IV in 250 ml D5W over 1 hr.
  IL-12 transduced TIL: On day 0 (one to four days after the last dose of fludarabine), cells will be infused intravenously (i.v.) on the Patient Care Unit over 20 to 30 minutes.
Period: Phase 1-Dose Escalation-Cohorts 1-4
Arm/Group | Group 1 - CD8 + TIL Expressing IL-12 1x10^6 (Phase 1) | Group 2 - CD8 + TIL Expressing IL-12 3x10^6 (Phase 1) | Group 3 - CD8 + TIL Expressing IL-12 1x10^7 (Phase 1) | Group 4 - CD8 + TIL Expressing IL-12 3x10^7 (Phase 1) | Group 5 - Bulk TIL Expressing IL-12 1x10^7 (Phase 1) | Group 6 - Bulk TIL Expressing IL-12 3x10^7 (Phase 1) | Group 7- Bulk TIL Expressing IL-12 1x10^8 (Phase 1) | Group 8 - Bulk TIL Expressing IL-12 3x10^8 (Phase 1) | Group 9 - Bulk TIL Expressing IL-12 1x10^9 (Phase 1) | Group 10 - Bulk TIL Expressing IL12 3x10^9 (Phase 1) | Group 11 - Bulk TIL Expressing MTD 1x10^9 (Phase 2)
Started | 1 | 1 | 6 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 1 | 1 | 6 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 1-Dose Escalation-Cohorts 5-10
Arm/Group | Group 1 - CD8 + TIL Expressing IL-12 1x10^6 (Phase 1) | Group 2 - CD8 + TIL Expressing IL-12 3x10^6 (Phase 1) | Group 3 - CD8 + TIL Expressing IL-12 1x10^7 (Phase 1) | Group 4 - CD8 + TIL Expressing IL-12 3x10^7 (Phase 1) | Group 5 - Bulk TIL Expressing IL-12 1x10^7 (Phase 1) | Group 6 - Bulk TIL Expressing IL-12 3x10^7 (Phase 1) | Group 7- Bulk TIL Expressing IL-12 1x10^8 (Phase 1) | Group 8 - Bulk TIL Expressing IL-12 3x10^8 (Phase 1) | Group 9 - Bulk TIL Expressing IL-12 1x10^9 (Phase 1) | Group 10 - Bulk TIL Expressing IL12 3x10^9 (Phase 1) | Group 11 - Bulk TIL Expressing MTD 1x10^9 (Phase 2)
Started | 0 | 0 | 0 | 0 | 1 | 4 | 3 | 3 | 4 | 4 | 0
Completed | 0 | 0 | 0 | 0 | 1 | 4 | 2 | 3 | 2 | 3 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0
Not completed — Death during treatment | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Not completed — Not treated | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Period: Phase 2- MTD/Anti-IL-12 Cells-Cohort 11
Arm/Group | Group 1 - CD8 + TIL Expressing IL-12 1x10^6 (Phase 1) | Group 2 - CD8 + TIL Expressing IL-12 3x10^6 (Phase 1) | Group 3 - CD8 + TIL Expressing IL-12 1x10^7 (Phase 1) | Group 4 - CD8 + TIL Expressing IL-12 3x10^7 (Phase 1) | Group 5 - Bulk TIL Expressing IL-12 1x10^7 (Phase 1) | Group 6 - Bulk TIL Expressing IL-12 3x10^7 (Phase 1) | Group 7- Bulk TIL Expressing IL-12 1x10^8 (Phase 1) | Group 8 - Bulk TIL Expressing IL-12 3x10^8 (Phase 1) | Group 9 - Bulk TIL Expressing IL-12 1x10^9 (Phase 1) | Group 10 - Bulk TIL Expressing IL12 3x10^9 (Phase 1) | Group 11 - Bulk TIL Expressing MTD 1x10^9 (Phase 2)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Did not receive cells | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 - CD8 + TIL Expressing IL-12 1x10^6 (Phase 1) | Group 2 - CD8 + TIL Expressing IL-12 3x10^6 (Phase 1) | Group 3 - CD8 + TIL Expressing IL-12 1x10^7 (Phase 1) | Group 4 - CD8 + TIL Expressing IL-12 3x10^7 (Phase 1) | Group 5 - Bulk TIL Expressing IL-12 1x10^7 (Phase 1) | Group 6 - Bulk TIL Expressing IL-12 3x10^7 (Phase 1) | Group 7- Bulk TIL Expressing IL-12 1x10^8 (Phase 1) | Group 8 - Bulk TIL Expressing IL-12 3x10^8 (Phase 1) | Group 9 - Bulk TIL Expressing IL-12 1x10^9 (Phase 1) | Group 10 - Bulk TIL Expressing IL12 3x10^9 (Phase 1) | Group 11 - Bulk TIL Expressing MTD 1x10^9 (Phase 2) | Total
Number analyzed (Participants) | 1 | 1 | 6 | 1 | 1 | 4 | 3 | 3 | 4 | 4 | 6 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 6 | 1 | 1 | 4 | 3 | 3 | 3 | 3 | 5 | 31
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.0 (0) | 50.0 (0) | 39.0 (11.5) | 48.0 (0) | 60.0 (0) | 57.3 (10.9) | 49.0 (14.5) | 56.0 (9.6) | 53.5 (16.2) | 55.8 (12.2) | 49.3 (16.5) | 50.7 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 1 | 2 | 0 | 9
  Male | 0 | 1 | 5 | 1 | 1 | 3 | 1 | 2 | 3 | 2 | 6 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
  Not Hispanic or Latino | 1 | 1 | 6 | 1 | 1 | 4 | 3 | 2 | 4 | 3 | 6 | 32
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 1 | 1 | 6 | 1 | 1 | 4 | 3 | 3 | 4 | 3 | 6 | 33
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 6 | 1 | 1 | 4 | 3 | 3 | 4 | 4 | 6 | 34

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: The MTD was determined by evaluating dose limiting toxicities (DLT) of participants that received increasing doses of intravenous infusion of IL-12 gene transduced tumor infiltrating lymphocytes (TIL) (i.e., 1x10^6, 3x10^6, 3x10^7, 1x10^7, 3x10^7, 1x10^8, 3x10^8, 1x10^9, and 3x10^9) in cohorts 1-10. Maximum tolerated cell dose is the highest dose at which </= 1 of 6 patients experienced a DLT (i.e. grade 2 or greater allergic reaction)).
Time Frame: 4 years
Measure: Number; unit: Cells
Groups:
- All Phase I Participants: All phase I participants who received at least one dose intravenously of CD8 + TIL expressing IL-12 in Groups 1-4, and Bulk TIL expressing IL-12 in Groups 5-10 (i.e., CD8 + TIL expressing IL-12 1x10^6, CD8 + TIL expressing IL-12 3x10^6, CD8 + TIL expressing IL-12 3x10^7, CD8 + TIL expressing IL-12 3x10^7, Bulk TIL expressing IL-12 1x10^7, Bulk TIL expressing IL-12 3x10^7, Bulk TIL expressing IL-12 1x10^8, Bulk TIL expressing IL-12 3x10^8, Bulk TIL expressing IL-12 1x10^9, and Bulk TIL expressing IL-12 3x10^9) respectively.
Arm/Group | All Phase I Participants
Number analyzed (Participants) | 28
Cells | 1,000,000,000

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For a detailed list of adverse events, see the adverse event module.
Time Frame: 49 months and 20 days
Measure: Number; unit: participants
Arm/Group | Group 1 - CD8 + TIL Expressing IL-12 1x10^6 (Phase 1) | Group 2 - CD8 + TIL Expressing IL-12 3x10^6 (Phase 1) | Group 3 - CD8 + TIL Expressing IL-12 1x10^7 (Phase 1) | Group 4 - CD8 + TIL Expressing IL-12 3x10^7 (Phase 1) | Group 5 - Bulk TIL Expressing IL-12 1x10^7 (Phase 1) | Group 6 - Bulk TIL Expressing IL-12 3x10^7 (Phase 1) | Group 7- Bulk TIL Expressing IL-12 1x10^8 (Phase 1) | Group 8 - Bulk TIL Expressing IL-12 3x10^8 (Phase 1) | Group 9 - Bulk TIL Expressing IL-12 1x10^9 (Phase 1) | Group 10 - Bulk TIL Expressing IL12 3x10^9 (Phase 1) | Group 11 - Bulk TIL Expressing MTD 1x10^9 (Phase 2)
Number analyzed (Participants) | 1 | 1 | 6 | 1 | 1 | 4 | 3 | 3 | 4 | 4 | 6
participants | 1 | 1 | 6 | 1 | 1 | 4 | 3 | 3 | 4 | 4 | 6

3. Primary Outcome: Response (Complete Response (CR) + Partial Response (PR)) to Therapy
Description: Response was determined by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.0. Complete response (CR) is disappearance of all target lesions. Partial response (PR) is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions taking as reference the baseline um LD. Progressive disease (PD) is at least a 20% increase in the sum of LD of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more lesions.
Time Frame: 4 years
Measure: Number; unit: participants
Arm/Group | Group 1 - CD8 + TIL Expressing IL-12 1x10^6 (Phase 1) | Group 2 - CD8 + TIL Expressing IL-12 3x10^6 (Phase 1) | Group 3 - CD8 + TIL Expressing IL-12 1x10^7 (Phase 1) | Group 4 - CD8 + TIL Expressing IL-12 3x10^7 (Phase 1) | Group 5 - Bulk TIL Expressing IL-12 1x10^7 (Phase 1) | Group 6 - Bulk TIL Expressing IL-12 3x10^7 (Phase 1) | Group 7- Bulk TIL Expressing IL-12 1x10^8 (Phase 1) | Group 8 - Bulk TIL Expressing IL-12 3x10^8 (Phase 1) | Group 9 - Bulk TIL Expressing IL-12 1x10^9 (Phase 1) | Group 10 - Bulk TIL Expressing IL12 3x10^9 (Phase 1) | Group 11 - Bulk TIL Expressing MTD 1x10^9 (Phase 2)
Number analyzed (Participants) | 1 | 1 | 6 | 1 | 1 | 4 | 3 | 3 | 4 | 4 | 6
participants
  Complete Response (CR) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Partial Response (PR) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1
  Progressive Disease (PD) | 1 | 1 | 6 | 0 | 1 | 4 | 2 | 2 | 2 | 0 | 3
  Not Assessed (NA) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 1
  Not Evaluable (NE) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Arm/Group | Group 1 - CD8 + TIL Expressing IL-12 1x10^6 (Phase 1) | Group 2 - CD8 + TIL Expressing IL-12 3x10^6 (Phase 1) | Group 3 - CD8 + TIL Expressing IL-12 1x10^7 (Phase 1) | Group 4 - CD8 + TIL Expressing IL-12 3x10^7 (Phase 1) | Group 5 - Bulk TIL Expressing IL-12 1x10^7 (Phase 1) | Group 6 - Bulk TIL Expressing IL-12 3x10^7 (Phase 1) | Group 7- Bulk TIL Expressing IL-12 1x10^8 (Phase 1) | Group 8 - Bulk TIL Expressing IL-12 3x10^8 (Phase 1) | Group 9 - Bulk TIL Expressing IL-12 1x10^9 (Phase 1) | Group 10 - Bulk TIL Expressing IL12 3x10^9 (Phase 1) | Group 11 - Bulk TIL Expressing MTD 1x10^9 (Phase 2)
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 2/6 | 0/1 | 0/1 | 0/4 | 1/3 | 1/3 | 1/4 | 1/4 | 2/6
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 6/6 | 1/1 | 1/1 | 4/4 | 3/3 | 3/3 | 4/4 | 4/4 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 - CD8 + TIL Expressing IL-12 1x10^6 (Phase 1) (N=1) | Group 2 - CD8 + TIL Expressing IL-12 3x10^6 (Phase 1) (N=1) | Group 3 - CD8 + TIL Expressing IL-12 1x10^7 (Phase 1) (N=6) | Group 4 - CD8 + TIL Expressing IL-12 3x10^7 (Phase 1) (N=1) | Group 5 - Bulk TIL Expressing IL-12 1x10^7 (Phase 1) (N=1) | Group 6 - Bulk TIL Expressing IL-12 3x10^7 (Phase 1) (N=4) | Group 7- Bulk TIL Expressing IL-12 1x10^8 (Phase 1) (N=3) | Group 8 - Bulk TIL Expressing IL-12 3x10^8 (Phase 1) (N=3) | Group 9 - Bulk TIL Expressing IL-12 1x10^9 (Phase 1) (N=4) | Group 10 - Bulk TIL Expressing IL12 3x10^9 (Phase 1) (N=4) | Group 11 - Bulk TIL Expressing MTD 1x10^9 (Phase 2) (N=6)
Platelets (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0x10e9/L) (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemoglobin (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombosis/thrombus/embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bilirubin (Hyperbilirubinemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Creatinine (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombotic microangiopathy (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — (e.g., thrombotic thrombocytopenic purpura (TTP) or hemolytic uremic syndrome (HUS)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
AST, SGOT (serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 - CD8 + TIL Expressing IL-12 1x10^6 (Phase 1) (N=1) | Group 2 - CD8 + TIL Expressing IL-12 3x10^6 (Phase 1) (N=1) | Group 3 - CD8 + TIL Expressing IL-12 1x10^7 (Phase 1) (N=6) | Group 4 - CD8 + TIL Expressing IL-12 3x10^7 (Phase 1) (N=1) | Group 5 - Bulk TIL Expressing IL-12 1x10^7 (Phase 1) (N=1) | Group 6 - Bulk TIL Expressing IL-12 3x10^7 (Phase 1) (N=4) | Group 7- Bulk TIL Expressing IL-12 1x10^8 (Phase 1) (N=3) | Group 8 - Bulk TIL Expressing IL-12 3x10^8 (Phase 1) (N=3) | Group 9 - Bulk TIL Expressing IL-12 1x10^9 (Phase 1) (N=4) | Group 10 - Bulk TIL Expressing IL12 3x10^9 (Phase 1) (N=4) | Group 11 - Bulk TIL Expressing MTD 1x10^9 (Phase 2) (N=6)
PTT (Partial Thromboplastin TIme) (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 4 (4) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 3 (3) | 1 (1) | 0 (0)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 6 (6) | 1 (1) | 1 (1) | 4 (4) | 2 (2) | 3 (3) | 4 (4) | 4 (4) | 3 (3)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 6 (6) | 1 (1) | 1 (1) | 4 (4) | 3 (3) | 3 (3) | 4 (4) | 4 (4) | 6 (6)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 6 (6) | 1 (1) | 1 (1) | 4 (4) | 3 (3) | 3 (3) | 4 (4) | 4 (4) | 6 (6)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 6 (6) | 1 (1) | 1 (1) | 4 (4) | 3 (3) | 3 (3) | 4 (4) | 3 (3) | 6 (6)
Platelets (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 5 (5) | 1 (1) | 1 (1) | 4 (4) | 2 (2) | 3 (3) | 4 (4) | 4 (4) | 6 (6)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 5 (5) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 3 (3) | 3 (3) | 4 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 4 (4) | 1 (1) | 1 (1) | 3 (3) | 3 (3) | 3 (3) | 4 (4) | 4 (4) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 3 (3) | 3 (3) | 3 (3) | 3 (3) | 1 (1) | 2 (2)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 6 (6) | 1 (1) | 1 (1) | 4 (4) | 3 (3) | 3 (3) | 4 (4) | 4 (4) | 1 (1)
Pain (General disorders) | 1 (1) | 1 (1) | 6 (6) | 1 (1) | 1 (1) | 4 (4) | 3 (3) | 3 (3) | 3 (3) | 4 (4) | 3 (3)
Coagulation-Other (thrombotic microangiopathy) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cytokine release syndrome/acute infusion reaction (Immune system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombosis/thrombus/embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage, pulmonary/upper respiratory (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular and nodal arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage, GU (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Pleural effusion (non-malignant) (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Death not associated with CTCAE term (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage, GI (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal -Other (bloating) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritis/itching (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver dysfunction/failure (clinical) (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Edema:limb (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Weight gain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hemorrhage, CNS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Confusion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mood alteration (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Psychosis (hallucinations/delusions) (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision-blurred vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vascular-Other (anasarca) (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 3 (3) | 3 (3) | 4 (4) | 2 (2)
Rigors/chills (General disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 3 (3) | 3 (3) | 1 (1)
Sweating (diaphoresis) (General disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Weight loss (General disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Flushing (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 3 (3) | 2 (2)
Mucositis/stomatitis (clinical exam) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Alkaline phosphatase (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 4 (4) | 2 (2) | 1 (1) | 3 (3) | 4 (4) | 2 (2)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Creatinine (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuropathy:sensory (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pericardial effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 5 (5) | 1 (1) | 1 (1) | 4 (4) | 3 (3) | 3 (3) | 3 (3) | 2 (2) | 1 (1)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 6 (6) | 1 (1) | 1 (1) | 4 (4) | 3 (3) | 3 (3) | 2 (2) | 2 (2) | 0 (0)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 6 (6) | 1 (1) | 1 (1) | 4 (4) | 1 (1) | 3 (3) | 4 (4) | 3 (3) | 2 (2)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 3 (3) | 3 (3) | 1 (1) | 0 (0)
Anorexia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 6 (6) | 1 (1) | 1 (1) | 4 (4) | 3 (3) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Febrile neutropenia (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 3 (3) | 4 (4) | 4 (4) | 5 (5) — (fever of unknown origin without clinically or microbiologically documented infection) (ANC <1.0x10e9/L, fever >=38.5 degrees C)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
AST, SGOT (serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 4 (4) | 1 (1) | 2 (2) | 4 (4) | 4 (4) | 2 (2)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 1 (1) | 4 (4) | 2 (2) | 2 (2) | 4 (4) | 4 (4) | 3 (3)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain-Other (generalized pain) (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to the unexpected toxicities, likely attributable to the tumor infiltrating lymphocytes (TIL) transduced with IL-12, and low percentage of durable responses, we decided to close this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No